CLINICAL TRIAL: NCT03513861
Title: Family Assisted Severe Febrile Illness Therapy (FASTER) for Critically-ill Kenyan Children
Brief Title: Family Assisted Severe Febrile Illness Therapy for Critically-ill Kenyan Children
Acronym: FASTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Amelie von Saint Andre-von Arnim, Assistant Professor, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 24080017
Record Dates: First submitted 2018-01-06; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Febrile Illness
Keywords: Low and Middle Income Countries; Limited resource settings; Early warning signs
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim 1: Parental FASTER tool training (Experimental): The goal is to see whether the child's parent/ guardian can be trained in overall severity of illness assessment using the FASTER Tool, to match the performance of a professional.
  Interventions: Other: FASTER Assessment tool
- Aim 2: Intervention group (Active Comparator): The intervention group parents will be taught the FASTER assessment tool. Intervention group parents will each be asked to monitor their own hospitalized child hourly using the FASTER assessment tool, and put up color-coded flags indicating severity of illness to the healthcare team. Parents will record the frequency of healthcare provider assessments of their child over the 24 hour intervention period.
  Interventions: Other: FASTER Assessment tool
- Aim 2: Control Group (No Intervention): The control group parents will not be taught the FASTER assessment tool. Hence they will not be involved in monitoring their child, nor signaling severity of their child's illness per color-coded flag system. Control group parents will record the frequency of healthcare provider assessments of their child over the 24 hrs enrollment period.

INTERVENTIONS:
Other: FASTER Assessment tool — The FASTER assessment tool consists of monitoring mental status, respiratory distress and capillary refill time by parents of children admitted to the hospital with febrile illness. Parents in the intervention group are asked to monitor their child hourly with the FASTER tool and signal severity of illness to the healthcare team via color coded flag system. Number of healthcare provider - patient reassessments will be compared in intervention and control group.
  Arms: Aim 1: Parental FASTER tool training; Aim 2: Intervention group

SUMMARY:
The purpose of this pilot study is to improve inpatient monitoring of severely-ill children admitted to the hospital in low resource settings at Kenyatta National Hospital in Nairobi, Kenya. Given the high ratio of patients to medical staff in these settings, the lack of reliable patient monitoring tools, and the high rate of early inpatient mortality, we will prospectively train parents as monitoring aids of their hospitalized children. Early recognition and intervention in critical illness is important to avoid (further) organ failure. Parents will be taught how to assess their child's mental status, work of breathing and capillary refill time which will inform a 3-point severity of illness scale. The severity of illness will be conveyed by the parents to the medical staff via color-coded flag system. The goal is to increase the healthcare provider patient reassessment rate according to patients' level of severity to assist in early recognition and treatment of patients' deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Kenyatta National Hospital with severe febrile illness which includes presumed malaria, sepsis or septic shock, pneumonia, meningitis or encephalitis
* Available adult caregiver
* Enrollment within the first 8 hours of admission to the pediatric ward (modified to 16 hrs later)

Exclusion Criteria:

* Primary cause of admission is major bleed or hemorrhagic shock, severe trauma or burn, major surgery, known congenital heart disease
* Previous study enrollment
* No available adult caregiver
* Caregiver unable to give informed consent
* Caregiver not proficient in English or Swahili

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Healthcare provider assessment rate of patient | First 24 hrs after enrollment
  Number of assessments of study patient by nurses or doctors within the 24 hrs intervention period

SECONDARY OUTCOMES:
Association of number of healthcare provider assessments within 24 hours with survival to discharge. | First 24 hrs after enrollment
  Number of healthcare provider assessments will be associated with survival to discharge.
Association of number of healthcare provider assessments within 24 hours with hospital length of stay. | First 24 hrs after enrollment
  Number of healthcare provider assessments will be associated with hospital length of stay.
Association of number of healthcare provider assessments within 24 hours with need of patient transfer to the pediatric ICU (PICU). | First 24 hrs after enrollment
  Number of healthcare provider assessments will be associated with need for transfer to the PICU.
Association of number of healthcare provider assessments within 24 hours with need of patient transfer from the acute room to the regular pediatric ward. | First 24 hrs after enrollment
  Number of healthcare provider assessments will be associated with need for patient transfer from the acute room that provides closer monitoring to regular pediatric ward.
Association of number of healthcare provider assessments within 24 hours with number of clinical procedures and interventions performed. | First 24 hrs after enrollment
  Number of healthcare provider assessments will be associated with the number of clinical procedures performed on patients. Invasive clinical procedures include, but are not limited to lumbar puncture, thoracentesis, abscess drainage). Interventions included are blood transfusion given; antibiotics or antimalarials given; fluid bolus given.
Association of number of healthcare provider assessments within 24 hours with the change in Pediatric Early Warning Score (PEWS) between time of enrollment and 24 hour time point | First 24 hrs after enrollment
  Number of healthcare provider assessments will be associated with the change in patients' PEWS score between time of enrollment and 24 hrs status post enrollment. The bedside PEWS is measured by 6 components, including heart rate, systolic blood pressure, capillary refill time, respiratory rate, oxygen saturation, respiratory effort and oxygen therapy. The score ranges between zero to 24 point, with 24 point representing the highest severity level.
Initial PEWS and change in PEWS from enrollment to 24 hrs in intervention vs control group will be correlated with the need for patients requiring transfer to PICU. | First 24 hrs after enrollment
  The goal of this outcome is to see if patients with equivalent levels of illness severity in both intervention and control group, exhibit differences in need for transfer to the intensive care unit.
Initial PEWS and change in PEWS score over 24 hrs in intervention vs control group will be correlated with mortality. | First 24 hrs after enrollment
  The goal of this outcome is to see if patients with equivalent levels of illness severity in both intervention and control group, exhibit differences in mortality.
Proportion of concordant FASTER assessments between parents and research team for Aim 1 patients and Aim 2 intervention group patients | First 24 hrs after enrollment
  The goal of this outcome is to assess the accuracy of the parental FASTER assessments compared to the gold standard which is the research team's FASTER assessment.
Correlation of PEWS score with Research team's FASTER tool assessments for Aim 1 patients and in both control and intervention group for Aim 2 patients | First 24 hrs after enrollment
  The bedside PEWS is measured by 6 components, including heart rate, systolic blood pressure, capillary refill time, respiratory rate, oxygen saturation, respiratory effort and oxygen therapy. The score ranges between zero to 24 point, with 24 point representing the highest severity level.
Association of parental level of education with correct parental severity of illness level assessment compared to research team assessments in intervention group patients. | First 24 hrs after enrollment
  This outcome will assess if level of parental education has an impact on the correct use of the FASTER tool. There are up to 24 separate parental FASTER assessments and 4 research team assessments per patient. Parental and research team assessment have to occur within 1 hr of one another to qualify for comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Kenyatta National Hospital, Nairobi, Kenya

REFERENCES:
- [Derived] von Saint Andre-von Arnim AO, Kumar RK, Clark JD, Wilfond BS, Nguyen QP, Mutonga DM, Zimmerman JJ, Oron AP, Walson JL. Family-Assisted Severity of Illness Monitoring for Hospitalized Children in Low-Resource Settings-A Two-Arm Interventional Feasibility Study. Front Pediatr. 2022 May 23;10:804346. doi: 10.3389/fped.2022.804346. eCollection 2022. PMID 35676898
- [Derived] von Saint Andre-von Arnim AO, Kumar RK, Oron AP, Nguyen QP, Mutonga DM, Zimmerman J, Walson JL. Feasibility of Family-Assisted Severity of Illness Monitoring for Hospitalized Children in Low-Income Settings. Pediatr Crit Care Med. 2021 Feb 1;22(2):e115-e124. doi: 10.1097/PCC.0000000000002582. PMID 33031354